CLINICAL TRIAL: NCT02033694
Title: The Lipid-Rich Plaque (LRP) Study
Brief Title: The Lipid-Rich Plaque Study
Acronym: LRP
Status: Completed | Type: Observational
Sponsor: Infraredx (Industry)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: The LRP Study
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Lipid; Vulnerable Plaque; Plaque; Cholesterol; Near Infrared Spectroscopy; NIRS-IVUS; Intravascular Ultrasound; Angiography; Coronary Imaging
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Participants With 2 Years Follow up: Participants with NIRS-IVUS imaging at baseline and assigned to follow up for Non-Index Culprit Lesion related Major Adverse Cardiac Events (NC-MACE) for 2 years
  Interventions: Device: NIRS-IVUS Imaging (TVC Imaging System)

INTERVENTIONS:
Device: NIRS-IVUS Imaging (TVC Imaging System) — Diagnostic Imaging Catheter

SUMMARY:
The purpose of this study is to enhance medical knowledge of the causes of future coronary problems. Many studies in patients who have already experienced a coronary problem point to the danger associated with plaques that are rich in cholesterol. This study determines if the near-infrared method of detection of these fatty plaques can predict future events. If dangerous plaques can be identified, there are many treatments already available that could be tested for their ability to prevent coronary events.

ELIGIBILITY:
General Inclusion Criteria:

* Subjects presenting for coronary angiography in whom IVUS imaging is likely to be performed for clinical purposes.
* Greater than 18 years of age.
* Clinical presenting symptoms meeting one of the three criteria below:

  1. Subjects presenting with an acute coronary syndrome (ACS) including at least one of the following:

     1. Elevated cardiac biomarkers with CK-MB or troponin greater than upper limits of normal;
     2. ST depression or ST elevation >1mm in 2 or more contiguous leads in the absence of LVH, paced rhythm, BBB or early repolarization;
     3. A stabilized patient 24 to 72 hours post STEMI;
  2. Unstable angina pectoris;
  3. Stable angina pectoris and/or a positive functional study with evidence of ischemia.

Angiographic Inclusion Criteria

* At least one Suspected Index Culprit Lesion requiring imaging with IVUS and/or NIRS for clinical indications.
* At least two native epicardial coronary arteries (which may include the Suspected Index Culprit Artery) eligible for imaging with NIRS-IVUS.

IVUS/NIRS Imaging Inclusion Criterion

* A minimum of a total 50 mm of coronary artery not involved in a prior or Index Procedure PCI (including the 5mm borders on either edge of the site receiving PCI) must be scanned. This 50mm total length may include contributions from the Suspected Index Culprit Arteries and from Index Non-Culprit Arteries. This total length must include contributions from two or more native imaged arteries.

Exclusion Criteria:

* Unstable patients (STEMI within the prior 24 hours; cardiogenic shock, hypotension needing inotropes, hypoxia needing intubation, and IABP) and patients that had a procedural complication (coronary dissection, perforation or a complication that would necessitate immediate-unplanned revascularization) during index PCI procedure.
* History of CABG or planned CABG within 6 months following NIRS-IVUS imaging.
* Patient has additional lesion(s) that needs a staged PCI.
* Subject life expectancy is less than 2 years at time of index catheterization.
* Subject with ejection fraction (EF) <30%.
* Subject pacemaker dependent/paced rhythm.
* Subject pregnant and lactating.
* Any other factor that the investigator feels would put the patient at increased risk or otherwise make the patient unsuitable for participation in the protocol
* Patients undergoing performance of PCI in all three major vessels during the index PCI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting for coronary angiography in whom IVUS and/or NIRS evaluation is planned or could be utilized as part of their clinically-indicated evaluation will be screened for participation.
  All enrolled patients with a large LRP (Maximum Lipid Core Burden Index>250 in 4 mm or maxLCBI4mm>=250) was contacted by phone for each clinical follow up visit to determine if a new coronary event had occurred. A randomly selected half of the patients with a small, or no LRP (MaxLCBI4mm<250) received an identical follow-up. The remaining half of the small or no LRP group did not have follow up visits and therefore were not included in the primary analysis. The determination of the need for follow-up was made by a core lab and communicated to the clinical site.
Sampling Method: Non-Probability Sample
Enrollment: 1563 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — MedStar Heart Institute
Locations (41):
- United States (31):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Palmetto General Hospital, Hialeah, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Palm Beach Gardens Medical Center, Palm Beach Gardens, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Emory Midtwon, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Alexian Brothers Heart and Vascular Institute, Elk Grove Village, Illinois
  - St. John's Springfield, Springfield, Illinois
  - Community Heart & Vascular, Indianapolis, Indiana
  - Methodist, Merrillville, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - McLaren Bay Region, Bay City, Michigan
  - St. John's, Detroit, Michigan
  - McLaren-Macomb, Mount Clemens, Michigan
  - Crittenton Hospital, Rochester, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - LIJ Health System, New York, New York
  - New York Presbyterian Hospital Cornell, New York, New York
  - Metrohealth, Cleveland, Ohio
  - Hillcrest Oklahoma Heart Institute, Tulsa, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Heart Hospital Plano, Plano, Texas
  - Davis Hospital and Medical Center, Layton, Utah
  - Charleston Area Medical Center, Charleston, West Virginia
- San Biovanni Hospital, Rome, Italy
- Latvian Centre of Cardiology, Riga, Latvia
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - Radboud University Medical Centre, Nijmegen
  - Erasmus Medical Centre, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
- SUSCCH, a.s., Banská Bystrica, Slovakia
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank
  - University of Edinburgh, Edinburgh
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Waksman R, Torguson R, Spad MA, Garcia-Garcia H, Ware J, Wang R, Madden S, Shah P, Muller J. The Lipid-Rich Plaque Study of vulnerable plaques and vulnerable patients: Study design and rationale. Am Heart J. 2017 Oct;192:98-104. doi: 10.1016/j.ahj.2017.02.010. Epub 2017 Feb 16. PMID 28938968
- [Background] Waksman R, Di Mario C, Torguson R, Ali ZA, Singh V, Skinner WH, Artis AK, Cate TT, Powers E, Kim C, Regar E, Wong SC, Lewis S, Wykrzykowska J, Dube S, Kazziha S, van der Ent M, Shah P, Craig PE, Zou Q, Kolm P, Brewer HB, Garcia-Garcia HM; LRP Investigators. Identification of patients and plaques vulnerable to future coronary events with near-infrared spectroscopy intravascular ultrasound imaging: a prospective, cohort study. Lancet. 2019 Nov 2;394(10209):1629-1637. doi: 10.1016/S0140-6736(19)31794-5. Epub 2019 Sep 27. PMID 31570255
- [Derived] Torguson R, Mintz GS, Di Mario C, Ten Cate T, Ali ZA, Singh V, Skinner W, Zhang C, Shea C, Kuku KO, Garcia-Garcia HM, Waksman R. Disparities among Black and White patients in plaque burden and composition and long-term impact. Cardiovasc Revasc Med. 2023 Oct;55:28-32. doi: 10.1016/j.carrev.2023.04.023. Epub 2023 May 1. PMID 37271594
- [Derived] Case BC, Torguson R, Mintz GS, Di Mario C, Medranda GA, Zhang C, Shea C, Garcia-Garcia HM, Waksman R. Additive Effect of Multiple High-Risk Coronary Artery Segments on Patient Outcomes: LRP Study Sub-Analysis. Cardiovasc Revasc Med. 2023 Jan;46:38-43. doi: 10.1016/j.carrev.2022.08.008. Epub 2022 Aug 6. PMID 36058829
- [Derived] Torguson R, Mintz GS, Case BC, Di Mario C, Zhang C, Shea C, Garcia-Garcia HM, Waksman R. Correlation between lipidic content and arterial-wall plaque burden: A Lipid Rich Plaque study sub-analysis. Int J Cardiol. 2022 Nov 1;366:32-34. doi: 10.1016/j.ijcard.2022.07.024. Epub 2022 Jul 13. PMID 35842005
- [Derived] Case BC, Shea C, Torguson R, Zhang C, Yerasi C, Medranda GA, Kuku KO, Garcia-Garcia HM, Mintz GS, Waksman R. Impact of Baseline Imaging of Non-Culprit Coronary Lesions on Adverse Events: Insight From LRP Study. Cardiovasc Revasc Med. 2022 Jun;39:1-5. doi: 10.1016/j.carrev.2021.12.012. Epub 2021 Dec 13. PMID 34972665
- [Derived] Torguson R, Shlofmitz E, Mintz GS, Mario CD, Cate TT, Ali ZA, Singh V, Skinner W, Zhang C, Shea C, Garcia-Garcia HM, Waksman R. Frequency of Lipid-Rich Coronary Plaques in Stable Angina Pectoris versus Acute Coronary Syndrome (from the Lipid Rich Plaque Study). Am J Cardiol. 2021 Nov 1;158:1-5. doi: 10.1016/j.amjcard.2021.07.033. Epub 2021 Aug 28. PMID 34465457
- [Derived] Bambagioni G, Di Mario C, Torguson R, Demola P, Ali Z, Singh V, Skinner W, Artis A, Cate TT, Zhang C, Garcia-Garcia HM, Doros G, Mintz GS, Waksman R. Lipid-rich plaques detected by near-infrared spectroscopy predict coronary events irrespective of age: A Lipid Rich Plaque sub-study. Atherosclerosis. 2021 Oct;334:17-22. doi: 10.1016/j.atherosclerosis.2021.08.022. Epub 2021 Aug 14. PMID 34455112
- See also: The Lipid-Rich Plaque Study of vulnerable plaques and vulnerable patients: Study design and rationale. Am Heart J. 2017 — https://www.ncbi.nlm.nih.gov/pubmed/28938968
- See also: Identification of patients and plaques vulnerable to future coronary events with near-infrared spectroscopy intravascular ultrasound imaging: a prospective, cohort study. Lancet. 2019 — https://www.ncbi.nlm.nih.gov/pubmed/31570255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled patients with a large LRP (Maximum Lipid Core Burden Index>250 in 4 mm or maxLCBI4mm>=250) were assigned to 2 year follow up to determine if a new coronary event had occurred. A randomly selected half of the patients with a small or no LRP (MaxLCBI4mm<250) had 2 year follow up.
Pre-assignment Details: A randomly selected half of the patients with a small or no LRP (MaxLCBI4mm<250) did not have 2 year follow up and were not included in the primary analyses. This reduced the total number of patients followed for two years to 1271 patients.
Groups:
- Participants With 2 Year Follow up: Participants with NIRS-IVUS imaging at baseline and assigned to follow up for Non-Index Culprit Lesion related Major Adverse Cardiac Events (NC-MACE) for 2 years
Period: Overall Study
Arm/Group | Participants With 2 Year Follow up
Started | 1271
Completed | 1271
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With 2 Year Follow up
Number analyzed (Participants) | 1271
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 388
  Male | 883
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participant could identify as more than one race/ethnicity and may be counted in more than one race/ethnicity category
  Participants
    Caucasian | 942
    African American | 158
    Asian Pacific | 44
    Native American | 0
    Other | 128
    Hispanic | 101
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 187
  Latvia | 10
  United States | 1001
  United Kingdom | 46
  Italy | 10
  Slovakia | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Stratified as Non-Index Culprit Lesion Related Major Adverse Cardiac Events (NC-MACE) or No NC-MACE and Association With maxLCBI4mm as a Continuous Variable
Description: Association of maximum 4 mm Lipid Core Burden Index (maxLCBI4mm) as a continuous value in 100 unit increments in all imaged arteries and NC-MACE at both (1) Patient Level and (2) Plaque Level
  Non-Index Culprit Lesion related Major Adverse Cardiac Events (NC-MACE) is defined as a composite of:
  * cardiac death
  * cardiac arrest
  * non-fatal myocardial infarction (MI)
  * acute coronary syndrome
  * revascularization by coronary artery bypass graft (CABG) or percutaneous intervention (PCI)
  * rehospitalization for progressive angina, related to a non-index culprit lesion
Time Frame: 2 years
Population: Patients assigned to 2 year follow up were analyzed, at the patient and plaque level, to test the association between maximum 4 mm Lipid Core Burden Index (maxLCBI4mm) and Non-Index Culprit Lesion related Major Adverse Cardiac Events (NC-MACE).
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With 2 Year Follow up
Number analyzed (Participants) | 1271
Participants
  Participants with NC-MACE | 104
  Participants with No NC-MACE | 1167
Statistical Analysis 1: Comparison: Participants With 2 Year Follow up; Hypothesis 1 (Vulnerable Patient Hypothesis) first fit a univariate proportional hazards regression model in which maxLCBI4mm is the only independent variable and NC-MACE during 2 years is the outcome. The null hypothesis tested by the Wald test that the regression coefficient in a proportional hazards regression model is significantly different from 0. This analysis determined whether maxLCBI4mmI is a risk factor for NC-MACE; Test type: Other; p = 0.0004, Regression, Cox; Cox Proportional Hazard = 1.21, 95% CI 2-sided [1.09 to 1.35]
Statistical Analysis 2: Comparison: Participants With 2 Year Follow up; Hypothesis 2 (Vulnerable Plaque Hypothesis) first fit a univariate proportional hazards regression model in which maxLCBI4mm in the coronary artery segment is the measure of exposure and NC-MACE during 2 years caused by a new culprit lesion in that segment is the outcome. This analysis was performed with adjustment for the potential clustering effect within patient utilizing the Wei, Lin and Weissfeld (WLW) methodology. This analysis determined whether maxLCBI4mm is a risk factor NC-MACE; Test type: Other; p < 0.0001, Regression, Cox; Cox Proportional Hazard = 1.45, 95% CI 2-sided [1.30 to 1.60]

2. Secondary Outcome: Number of Participants Stratified as NC-MACE or No NC-MACE and Association With maxLCBI4mm More Than a Threshold of 400
Description: Association of maxLCBI4mm more than and less than a threshold of 400 in all imaged arteries and NC-MACE at both (1) Patient Level and (2) Plaque Level
  Non-Index Culprit Lesion related Major Adverse Cardiac Events (NC-MACE) is defined as a composite of:
  * cardiac death
  * cardiac arrest
  * non-fatal myocardial infarction (MI)
  * acute coronary syndrome
  * revascularization by coronary artery bypass graft (CABG) or percutaneous intervention (PCI)
  * rehospitalization for progressive angina, related to a non-index culprit lesion
Time Frame: 2 years
Population: Patients assigned to 2 year follow up were analyzed, at the patient and plaque level to test the association between maximum 4mm Lipid Core Burden index (maxLCBI4mm) >400 and Non-Index Culprit Lesion related Major Cardiac Events (NC-MACE)
Measure: Count of Participants; unit: Participants
Groups:
- Participants With 2 Year Follow up: Participants with NIRS-IVUS imaging at baseline and follow up for 2 years
Arm/Group | Participants With 2 Year Follow up
Number analyzed (Participants) | 1271
Participants
  Participants with NC-MACE | 104
  Participants with No NC-MACE | 1167
Statistical Analysis 1: Comparison: Participants With 2 Year Follow up; Secondary Hypothesis 1 (Vulnerable Patient)- Cox proportional hazards regression model to assess a threshold of maxLCBI4mm > 400 as the independent variable and NC-MACE during 2 years as the outcome; Test type: Other; p < 0.0001, Regression, Cox; Cox Proportional Hazard = 2.18, 95% CI 2-sided [1.48 to 3.22]
Statistical Analysis 2: Comparison: Participants With 2 Year Follow up; Secondary Hypothesis 2 (Vulnerable Plaque)- Cox proportional hazards regression model to assess a threshold of maxLCBI4mm > 400 in the coronary artery segment as the independent variable and NC-MACE during 2 years caused by a new culprit lesion in that segment is the outcome; Test type: Other; p < 0.0001, Regression, Cox; Cox Proportional Hazard = 4.22, 95% CI 2-sided [2.39 to 7.45]

ADVERSE EVENTS:
Time Frame: 2 years
Description: The device has been approved as safe for imaging of coronary arteries by the FDA. Experience in greater than 5,000 patients has shown that the device safety profile does not differ from that of a conventional IVUS catheter. Serious adverse events associated with the device in the additional, non-culprit vessels were collected because this was the additional requirement for the study outside of routine medical care.
Groups:
- All Patients With Baseline NIRS-IVUS Imaging: Participants with NIRS-IVUS imaging at baseline
Arm/Group | All Patients With Baseline NIRS-IVUS Imaging
All-Cause Mortality (participants affected / at risk) | 0/1563
Serious Adverse Events (participants affected / at risk) | 6/1563
Other Adverse Events (participants affected / at risk) | 0/1563
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients With Baseline NIRS-IVUS Imaging (N=1563)
Dissection (Cardiac disorders) | 4 (4) — Intraprocedural complication
Bradycardia (Cardiac disorders) | 1 (1) — Intraprocedural complication
Thrombus with Chest Pain (Cardiac disorders) | 1 (1) — Intraprocedural complication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT02033694/Prot_SAP_000.pdf